CLINICAL TRIAL: NCT00812331
Title: An Open-label Trial in Genotype 2, 3, 4, 5 and 6 Hepatitis C-infected Subjects to Evaluate the Antiviral Activity, Safety, Tolerability and Pharmacokinetics of TMC435350 Following 7 Days Once Daily Dosing as Monotherapy.
Brief Title: A Study to Assess the Anti-viral Activity, Safety, Tolerability and Pharmacokinetics of TMC435350 in Participants Infected With Hepatitis C-Virus (HCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012604; TMC435350-TiDP16-C202 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Genotype 2 (Experimental): Participants with chronic genotype 2 hepatitis C virus (HCV) infection
  Interventions: Drug: TMC435
- Genotype 3 (Experimental): Participants with chronic genotype 3 HCV infection
  Interventions: Drug: TMC435
- Genotype 4 (Experimental): Participants with chronic genotype 4 HCV infection
  Interventions: Drug: TMC435
- Genotype 5 (Experimental): Participants with chronic genotype 5 HCV infection
  Interventions: Drug: TMC435
- Genotype 6 (Experimental): Participants with chronic genotype 6 HCV infection
  Interventions: Drug: TMC435

INTERVENTIONS:
Drug: TMC435 — From Day 1 to Day 7 all participants will take 200 mg TMC435350 as a single medication orally (by mouth) once daily.

SUMMARY:
The purpose of this study is to assess anti-viral activity (inhibition of viral growth) of TMC435350 in genotype 2,3,4,5 and 6 hepatitis C virus infected participants who have never received treatment for their hepatitis C infection.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) study to assess the antiviral activity, safety, tolerability and pharmacokinetics (explores what the body does to the medication) of TMC435350 hereafter referred to as TMC435. Approximately 40 participants will be divided in 5 groups as per the genotype (8 participants each group). The study will include a screening phase (up to 6 weeks), treatment phase (7 days) and a follow-up phase (30-35 days after the last dose of study medication). Safety evaluations will include assessment of adverse events, clinical laboratory tests and cardiovascular safety.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented chronic genotype 2, 3, 4, 5 or 6 hepatitis C virus (HCV) infection
* Participants who have never received treatment for their HCV infection
* Participants with either no cirrhosis or up to Child Pugh A liver disease
* Participants with plasma HCV genotype level of more than or equal to 100, 000 IU/mL at screening

Exclusion Criteria:

* Evidence of Child Pugh B or C liver disease at screening, decompensated liver disease defined as prior or current history of ascities, hepatic encephalopathy, esophageal or gastric varices
* Participants with diagnosed or suspected hepatocellular carcinoma
* Participants coinfected with human immunodeficiency virus type 1 or 2, or hepatitis A or B virus infection or active tuberculosis at screening
* Participants with any active clinically significant disease, or medical history or physical examination or electrocardiogram findings during screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (10):
- Belgium (4):
  - Bruges
  - Brussels
  - Ghent
  - Leuven
- Germany (4):
  - Berlin
  - Frankfurt
  - Freiburg im Breisgau
  - Hanover
- Thailand (2):
  - Bangkok
  - Chiang Mai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 participants from 3 countries were enrolled and started treatment in the study (17 participants in Belgium, 12 participants in Germany, and 8 participants in Thailand).
Pre-assignment Details: A total of 48 participants were screened of which 11 participants were not treated with TMC435. A total of 37 participants received study medication.
Groups:
- Genotype 2: Participants with chronic genotype 2 HCV infection who received 200 mg TMC435 as a single oral (by mouth) dose once daily for 7 days
- Genotype 3: Participants with chronic genotype 3 HCV infection who received 200 mg TMC435 as a single oral (by mouth) dose once daily for 7 days
- Genotype 4: Participants with chronic genotype 4 HCV infection who received 200 mg TMC435 as a single oral (by mouth) dose once daily for 7 days
- Genotype 5: Participants with chronic genotype 5 HCV infection who received 200 mg TMC435 as a single oral (by mouth) dose once daily for 7 days
- Genotype 6: Participants with chronic genotype 6 HCV infection who received 200 mg TMC435 as a single oral (by mouth) dose once daily for 7 days
Period: Overall Study
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Started | 6 | 8 | 8 | 7 | 8
Completed | 5 | 8 | 8 | 7 | 8
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6 | Total
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8 | 37
Age, Continuous [Median (Full Range); unit: years] | 43 [27 to 61] | 42 [18 to 56] | 47 [26 to 55] | 65 [48 to 69] | 49 [30 to 53] | 48 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 4 | 2 | 18
  Male | 2 | 5 | 3 | 3 | 6 | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 5 | 7 | 6 | 7 | 0 | 25
  Asian | 0 | 1 | 0 | 0 | 8 | 9
  Black | 1 | 0 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in log10 Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels
Description: The table below shows the mean changes from baseline in HCV RNA values (log10 IU/mL) per genotype on Day 3 and Day 7 during the TMC435 treatment period.
Time Frame: Baseline, Day 3, and Day 7
Population: Intent-to-treat (ITT) population - all randomized participants who received at least 1 dose of study medication (TMC435).
Measure: Mean (Standard Error); unit: log10 IU/mL
Groups:
- Genotype 2: Participants with chronic genotype 2 HCV infection who received 200 mg TMC435 as a single oral ((by mouth) dose once daily for 7 days.
- Genotype 3: Participants with chronic genotype 3 HCV infection who received 200 mg TMC435 as a single oral ((by mouth) dose once daily for 7 days.
- Genotype 4: Participants with chronic genotype 4 HCV infection who received 200 mg TMC435 as a single oral ((by mouth) dose once daily for 7 days.
- Genotype 5: participants with chronic genotype 5 HCV infection who received 200 mg TMC435 as a single oral ((by mouth) dose once daily for 7 days.
- Genotype 6: participants with chronic genotype 6 HCV infection who received 200 mg TMC435 as a single oral ((by mouth) dose once daily for 7 days.
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
log10 IU/mL
  Day 3 | -2.02 (0.625) [-3.6 to -0.3] | 0.16 (0.263) [-0.7 to 1.8] | -3.43 (0.167) [-3.9 to -2.6] | -2.71 (0.335) [-4.0 to -1.5] | -3.57 (0.197) [-4.2 to -2.7]
  Day 7 | -2.46 (0.538) [-4.2 to -0.9] | -0.13 (0.175) [-1.0 to 0.6] | -3.66 (0.320) [-4.7 to -2.3] | -2.43 (0.357) [-3.2 to -0.7] | -4.40 (0.222) [-5.2 to -3.3]

2. Secondary Outcome: Number of Participants With a Decrease From Baseline of Greater Than or Equal to 2 log10 IU/mL in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) During the TMC435 Treatment Period
Description: The table below shows the number of participants with a decrease from baseline of greater than or equal to 2 log10 IU/mL in HCV RNA during the 7-day TMC435 treatment period.
Time Frame: Baseline, Day 3, Day 5 and Day 7
Population: Intent-to-treat (ITT) Population- all randomized subjects who received at least 1 dose of study medication (TMC435)
Measure: Number; unit: Participants
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
Participants
  Day 3 | 3 | 0 | 8 | 6 | 8
  Day 5 | 3 | 0 | 8 | 5 | 8
  Day 7 | 3 | 0 | 8 | 5 | 8

3. Secondary Outcome: Number of Participants With Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels Below the Limit of Quantification (Less Than 25 IU/mL) and Limit of Detection (Less Than 25 IU/mL Undetectable) During the TMC435 Treatment Period
Description: The table below shows the number of participants with plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels below limit of quantification (less than 25 IU/mL) and limit of detection (less than 25 IU/mL undetectable), respectively, during the 7-day TMC435 treatment period.
Time Frame: Baseline, Day 3, Day 5 and Day 7
Population: Intent-to-treat (ITT) Population - all randomized subjects who received at least 1 dose of study medication (TMC435)
Measure: Number; unit: Participants
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
Participants
  Day 3 (less than 25 IU/mL) | 0 | 0 | 0 | 0 | 0
  Day 3 (less than 25 IU/mL undetectable) | 0 | 0 | 0 | 0 | 0
  Day 5 (less than 25 IU/mL) | 0 | 0 | 2 | 0 | 1
  Day 5 (less than 25 IU/mL undetectable) | 0 | 0 | 1 | 0 | 0
  Day 7 (less than 25 IU/mL) | 0 | 0 | 3 | 0 | 1
  Day 7 (less than 25 IU/mL undetectable) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Who Experienced Viral Breakthrough During TMC435 Treatment Period
Description: The table below shows the number of participants who experienced viral breakthrough (defined as an increase greater than 1 log10 IU/mL in plasma level of hepatitis C virus [HCV] ribonucleic acid [RNA] from the lowest level reached, or a HCV RNA level greater than 100 IU/mL in participants who previously had HCV RNA levels undetectable [less than 25 IU/mL undetectable] or not quantifiable [less than 25 IU/mL detectable]) during the 7-day TMC435 treatment period.
Time Frame: During the 7-day of TMC435 treatment period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
Participants | 0 | 1 | 2 | 3 | 0

5. Secondary Outcome: Predose Plasma Concentration (C0h) of TMC435
Description: The table below shows the median predose plasma concentration (C0h) for all participants on Day 7 of the TMC435 treatment period.
Time Frame: Predose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
ng/mL | 3720 [164 to 8420] | 1310 [492 to 4220] | 6270 [1030 to 13100] | 4650 [80.1 to 14500] | 5440 [2280 to 11700]

6. Secondary Outcome: Minimum Plasma Concentration (Cmin) of TMC435
Description: The table below shows the median minimum plasma concentration (Cmin) for all participants on Day 7 of the TMC435 treatment period.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
ng/mL | 3320 [156 to 8420] | 1110 [463 to 3440] | 5450 [1030 to 13100] | 4230 [48.2 to 14300] | 4960 [2080 to 10600]

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of TMC435
Description: The table below shows the median maximum plasma concentration (Cmax) for all participants by genotype of hepatitis C virus infection on Day 7 of the TMC435 treatment period.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
ng/mL | 11250 [2360 to 18500] | 6580 [2760 to 13200] | 13500 [4530 to 26200] | 13600 [215 to 24700] | 14800 [3460 to 23000]

8. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of TMC435
Description: The table below shows the median time in hours for all participants (by genotype of hepatitis C virus infection) to reach the maximum plasma concentration (tmax) of TMC435 following treatment.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
hours | 4.01 [4.00 to 7.83] | 6.025 [4.02 to 10.08] | 6.04 [4.00 to 8.08] | 6.00 [4.00 to 8.02] | 6.00 [4.00 to 6.20]

9. Secondary Outcome: Average Steady-State Plasma Concentration (Css,av) of TMC435
Description: The table below shows the average steady-state TMC435 plasma concentration (Css,av) for all participants by genotype of hepatitis C virus infection on Day 7 during the TMC435 treatment period.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
ng/mL | 7115 [1110 to 12870] | 3081 [1410 to 7550] | 8843 [2954 to 20340] | 7850 [130.8 to 19660] | 9354 [2602 to 16180]

10. Secondary Outcome: Fluctuation Index (FI) of TMC435
Description: The table below shows the percentage of fluctuation (FI) (defined as the variation between maximum and minimum TMC435 plasma concentrations at steady-state) of TMC435 on Day 7 for participants by genotype of hepatitis C virus infection.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: % fluctuation
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
% fluctuation | 130.2 [78.35 to 210.4] | 149.4 [100.3 to 246.3] | 95.38 [56.77 to 161.1] | 93.12 [52.91 to 129.3] | 88.16 [53.04 to 127.6]

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration up to 24 Hours After Dosing (AUC24h) of TMC435
Description: The table below shows the area under the plasma concentration-time curve from the time of administration up to 24 hours after dosing (AUC24h) of TMC435 on Day 7 for all participants by genotype of hepatitis C virus infection.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: Intent-to-treat (ITT) population - as all randomized participants who received at least 1 dose of study medication (TMC435).
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
ng*h/mL | 170100 [26350 to 311000] | 74670 [34500 to 199500] | 212000 [70400 to 483000] | 189000 [3084 to 457600] | 227100 [63430 to 373500]

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time of Administration up to the Last Time Point With a Measurable Concentration After Dosing (AUClast) of TMC435
Description: The table below shows the area under the plasma concentration-time curve from time of administration up to the last time point with a measurable concentration after dosing (AUClast) on Day 7 for TMC435 by genotype of hepatitis C virus infection.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
ng*h/mL | 268000 [31400 to 712600] | 111500 [43680 to 272000] | 365500 [99320 to 1179000] | 360000 [3770 to 944400] | 411100 [117500 to 798900]

13. Secondary Outcome: Elimination Rate Constant of TMC435
Description: In the table below, median values for the elimination rate constant (the rate at which a drug is removed from the body expressed per unit of time, e.g., fraction/hour) for TMC435 are shown for participants by genotype of hepatitis C virus infection.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: 1/hour
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
1/hour | 0.05042 [0.01776 to 0.08666] | 0.06024 [0.04057 to 0.08552] | 0.04308 [0.01803 to 0.06955] | 0.03826 [0.03315 to 0.07737] | 0.03784 [0.01826 to 0.05926]

14. Secondary Outcome: Terminal Elimination Half-life (t1/2,Term) of TMC435
Description: The table below shows the terminal plasma half-life for TMC435 in participants analyzed by genotype of hepatitis C virus infection. The terminal plasma half-life of a drug is the time in hours required for the concentration of a drug in the body to fall to 50% after having reached a state of equilibrium following administration.
Time Frame: Predose, and at 0.5, 1, 2, 4, 6, 8, and 10 hours post-dose on Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5 | Genotype 6
Number analyzed (Participants) | 6 | 8 | 8 | 7 | 8
hours | 13.75 [7.998 to 39.04] | 11.51 [8.105 to 17.09] | 16.09 [9.966 to 38.44] | 18.12 [8.959 to 20.91] | 18.32 [11.70 to 37.95]

ADVERSE EVENTS:
Time Frame: From the date of signing of the Informed Consent Form onwards until 30-35 days after last TMC435 intake.
Description: 5% cutoff is restricted to Total group. Adverse events reported for the total group rather than by genotype because enrollment numbers by genotype were small.
Groups:
- Total: Participants with chronic genotype 2,3,4,5 or 6 HCV infection who received 200 mg TMC435 as a single oral (by mouth) dose once daily for 7 days
Arm/Group | Total
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 22/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=37)
Ileitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=37)
Influenza like illness (General disorders) | 9
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Lip swelling (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 3
Palpitations (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days